CLINICAL TRIAL: NCT04044859
Title: A Phase 1 Dose Escalation Study To Assess Safety And Efficacy Of ADP-A2M4CD8 As Monotherapy Or In Combination With Either Nivolumab Or Pembrolizumab In HLA-A2+ Subjects With MAGE-A4 Positive Tumors (SURPASS)
Brief Title: ADP-A2M4CD8 as Monotherapy or in Combination With Either Nivolumab or Pembrolizumab in HLA-A2+ Subjects With MAGE-A4 Positive Tumors (SURPASS)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: USWM CT, LLC (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0055-001
Record Dates: First submitted 2019-07-03; First posted 2019-08-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer; Esophageal Cancer; Esophagogastric Junction (EGJ); Gastric (Stomach) Cancer; Head and Neck Cancer; Melanoma; Ovarian Cancer; Non-small Cell Lung (NSCLC); Urothelial Cancer
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; MAGE-A4; Immuno-oncology; Metastatic; Urothelial; Head and Neck; Gastric (stomach); Esophagogastric Junction (EGJ); Non-small Cell Lung (NSCLC); Esophageal Cancer; Ovarian Cancer; Endometrial Cancer; Melanoma
MeSH Terms: conditions — Endometrial Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Melanoma; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified ADP-A2M4CD8 cells (Experimental)
  Interventions: Genetic: Autologous genetically modified ADP-A2M4CD8 cells alone or in combination with nivolumab every four weeks or pembrolizumab every 6 weeks

INTERVENTIONS:
Genetic: Autologous genetically modified ADP-A2M4CD8 cells alone or in combination with nivolumab every four weeks or pembrolizumab every 6 weeks — Infusion of autologous genetically modified ADP-A2M4CD8 on Day 1 alone or in combination with either nivolumab 480 mg IV every four weeks or pembrolizumab 400mg IV every 6 weeks

SUMMARY:
This study will investigate the safety and tolerability of ADP-A2M4CD8 T-cell therapy in subjects who have the appropriate human leukocyte antigen (HLA) and MAGE-A4 tumor antigen. Tumor indications include endometrial, esophageal, esophagogastric junction (EGJ), gastric, head and neck, melanoma, non-small cell lung (NSCLC), ovarian or urothelial cancer.

DETAILED DESCRIPTION:
Conditions:

Endometrial Esophageal Cancer Esophagogastric Junction (EGJ) Gastric (stomach) Head and Neck Melanoma Non-small Cell Lung (NSCLC) Ovarian Cancer

ELIGIBILITY:
* Key Inclusion criteria
* Age ≥18 and ≤ 75 years
* Subject is positive for at least 1 HLA-A*02 inclusion allele
* Histologically or cytogenetically confirmed diagnosis of urothelial cancer, esophageal, esophagogastric junction (EGJ) cancer, gastric cancer, non-small cell lung carcinoma (NSCLC), head and neck or ovarian cancer, endometrial cancer, melanoma
* Measurable disease according to RECIST v1.1 prior to leukapheresis and lymphodepletion.
* Tumor shows MAGE-A4 expression as confirmed by central laboratory
* ECOG Performance Status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥50% or the institutional lower limit of normal range, whichever is lower Note: other protocol defined Inclusion/Exclusion criteria may apply
* Subjects must have ≥ 90% room air oxygen saturation at rest at Screening (within 7 days of leukapheresis) and at Baseline.

Key exclusion criteria

* Positive for any HLA-A*02 allele other than: one of the inclusion alleles
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study
* Active autoimmune or immune mediated disease
* Leptomeningeal disease, carcinomatous meningitis or symptomatic CNS metastases
* Other prior malignancy that is not considered by the Investigator to be in complete remission. Clinically significant cardiovascular disease
* Uncontrolled intercurrent illness
* Active infection with human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or human T cell leukemia virus
* Pregnant or breastfeeding

Note: other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2037-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab | 2.5 years
  Determination of incidence of dose-limiting toxicities, adverse events and tolerable dose
To evaluate safety of ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab | Up to 15 years
  Incidence of patients with Replication-competent Retrovirus, persistence of ADP-A2M4CD8 T-cells and incidence of insertional oncogenesis.

SECONDARY OUTCOMES:
Anti-tumour activity: Overall Response Rate (ORR) | 2.5 years
  ORR is defined as incidence of complete responses or partial responses as assessed by RECIST v1.1
Anti-tumor activity: Best overall response (BOR) | 2.5 years
  BOR is per RECIST V1.1.
Time to response (TTR) | 2.5 years
  For patients who are observed to respond to ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab, the time taken to achieve a partial response or complete response (TTR) is assessed.
Duration of Response (DOR) | 2.5 years
  For patients who are observed to respond to ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab, the DOR is the date of first response (including confirmation) up until disease progression per RECIST v 1.1 or death
Duration of stable disease (DoSD) | 2.5 years
  For patients who are observed to have stable disease by RECIST v 1.1, the duration of period of stable disease until disease progression or death
Progression Free Survival (PFS) | 2.5 years
  PFS is assessed from date of infusion of ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab up until the date of disease progression per RECIST v1.1 or death.
Overall Survival (OS) | 15 years
  OS is assessed from date of infusion of ADP-A2M4CD8 as monotherapy or in combination with either nivolumab or pembrolizumab up until the date of patient death.

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (17):
- United States (9):
  - Name of Institution: Orlando Health Cancer Institute, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University - School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Duke Cancer Institute, Durham, North Carolina
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (7):
  - Hospital Universitario 12 De Octubre, Madrid, Avenida de Cordoba S/n
  - Clinica Universitaria de Navarra, Pío, Pamplona
  - Hospital Clinico de Valencia, Ibanez, Valencia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio, Seville